CLINICAL TRIAL: NCT06626360
Title: SCreening fOr Malnutrition and Obesity in Patients With COVID-19 and Other Diseases
Brief Title: Screening for Malnutrition in Obese Patients
Acronym: SCOOP
Status: Recruiting | Type: Observational
Sponsor: HAN University of Applied Sciences (Other)
Collaborators: Amsterdam University of Applied Sciences (Other); National Institute for Public Health and the Environment (RIVM) (Other Government); Erasmus Medical Center (Other); Wageningen University and Research (Other); Gelderse Vallei Hospital (Other); Amsterdam UMC, location VUmc (Other); Amsterdam UMC, location AMC (Other)
Responsible Party: Principal Investigator, dr. Marian de van der Schueren, Professor of Nutrition, Dietetics and Lifestyle, HAN University of Applied Sciences
Other Study IDs: SCOOP; 6496655 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Overweight and Obese Adults; Malnutrition or Risk of Malnutrition
Keywords: Overweight; Obesity; Malnutrition
MeSH Terms: conditions — Overweight; Malnutrition; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with overweight or obesity: Inclusion criteria:
  * Age 18 years or older
  * Overweight (BMI of 25 kg/m² or higher)
  Exclusion criteria:
  * Physically or mentally unable to participate.
  * Severe cognitive disorder or severe emotional instability, as assessed by the attending nurse or physician.
  * Insufficient proficiency in the Dutch language to express themselves properly and no interpreter or assistant to help.
  * Patient resides in a nursing or care home.

SUMMARY:
More than half of the Dutch population is overweight or obese, which is associated with an increased risk of COVID-19 and worse outcomes during a COVID-19 infection. In addition, malnutrition and loss of muscle mass are often reported with COVID-19, as well as with cancer and other diseases. Malnutrition and overweight or obesity can coexist, even within the same individual. It is still unclear which mechanisms contribute to the worse outcomes of COVID-19 and other diseases in case of overweight, malnutrition, and a combination of both. The aim of this study is to identify which parameters are associated with worse disease outcomes through literature research and database research (COVID-19 and cancer, more than 150.000 participants). In addition, a clinical study will be conducted aiming to develop a simple screening tool for the recognition of the coexistence of malnutrition and overweight or obesity in clinical practice.

DETAILED DESCRIPTION:
Overweight and malnutrition are both common and have a significant societal impact as well as a negative effect on healthcare. They can also coexist, and may potentially reinforce each other. How the combination of both influences the course of COVID-19 and other diseases is still largely unknown. There is no simple set of parameters yet available to screen for the simultaneous occurrence of overweight and malnutrition.

This project has the following objectives:

* To evaluate the nutritional status (malnutrition, overweight, and the combination of both) and the (dietary) treatment of patients with COVID-19 in primary care (WP1).
* To assess the influence of various parameters of malnutrition and overweight and their effects on the outcomes of COVID-19 and cancer based on literature and data from existing Dutch cohorts (WP2 and WP3).

Based on this, to develop a screening tool for malnutrition in overweight; (WP4).

- Dissemination of the results (WP5).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Overweight (BMI of 25 kg/m² or higher)

Exclusion Criteria:

* Physically or mentally unable to participate.
* Severe cognitive disorder or severe emotional instability, as assessed by the attending nurse or physician.
* Insufficient proficiency in the Dutch language to express themselves properly and no interpreter or assistant to help.
* Patient resides in a nursing or care home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital in- and outpatients with overweight or obesity
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Malnutrition | 9 months
  Malnutrition will be assessed by a working definition based on the GLIM-criteria and a Delphi-study

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - OLVG, Amsterdam
  - Ziekenhuis Gelderse Vallei, Ede
  - ErasmusMC, Rotterdam

IPD SHARING:
Plan to Share IPD: No
Data first need to be analysed and published